CLINICAL TRIAL: NCT03884790
Title: A Pre-market, Multi-center, International, Open-label, Single-arm Study to Evaluate the Safety and Performance of a Class III Medical Device (GreenBone Implant) for Surgical Repair of Long Bone Defects
Brief Title: Pre-market Study to Evaluate Safety and Performance of GreenBone Implant (Long Bone Study)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The enrolment phase was halted prematurely due to logistic issues ( SARS-CoV2 pandemic). All patients enrolled completed the follow-up visits according to the study protocol.
Sponsor: GreenBone Ortho S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GB-02-18
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2024-06

CONDITIONS: Bone Substitutes; Bone Defect
Keywords: Bone substitute; Bone regeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical repair of long bone defects (Experimental): The Patients in the study group will be surgically treated and the GreenBone Bone Substitute will be implanted
  Interventions: Device: surgical repair of long bone defects

INTERVENTIONS:
Device: surgical repair of long bone defects — Current treatment of bone defects usually implies the use of bone grafts and/or biocompatible materials, to create a scaffold that bridges the defect, favoring the migration of cells from the neighboring tissues to fill the gap. Autograft and Allograft are the treatments most currently used for large bone loss, but both treatments have significant disadvantages. Different types of synthetic materials have been tested for repair of long bone gaps.
  However, at the moment, there is not any bone substitute with the ideal/desirable osteoinductive, osteoconductive and mechanical properties. GreenBone Implant is a synthetic, acellular, reabsorbable, new generation bone graft, being suitable for surgical reconstruction of bone defects.

SUMMARY:
Multi-center, international, prospective, open-label, single-arm, first-in-human clinical investigation. The Patients enrolled in this clinical investigation will undergo a scheduled surgery for the treatment of long bone defects up to 6 cm using GreenBone Implant. After the surgery, the Patients will be monitored at pre-scheduled visits up to 12 months. Adverse events, pain, quality of life and functional parameters, as well as X-ray and CT scan, will be evaluated at scheduled follow-up visits. An independent Data Safety Monitoring Board (DSMB) will review the safety reports at regular intervals and Serious Adverse Events (SAE) as soon as reported, to protect Patients participating in the study. The initial phase of the study contemplates the treatment of bone defects up to 3 cm. An adaptive interim analysis will be performed when the first 7 Patients will have completed the 6-month follow-up visit. The DSMB will review the results of the interim analysis with respect to the primary endpoint (safety), and provide one of the following recommendations to the Sponsor: a) to stop the study for unacceptable frequency and severity of adverse events or b) to continue the study up to 25 Patients recruited and to include at least 5 Patients with a longer bone defect (> 3 cm up to 6 cm).

DETAILED DESCRIPTION:
This is a pre-market multi-centre, international, open label, single-arm, study to evaluate the safety and performance of a Class III medical device (GreenBone Implant) for the treatment of long bone defect. Bone defects can result from malformation, high-energy traumatic events, bone resection due to different pathologies such as tumors or infections, or from the treatment of complex non-unions. Current treatment of bone defects usually implies the use of bone grafts and/or biocompatible materials, to create a scaffold that bridges the defect. Autograft and Allograft are the treatments most currently used for large bone loss, but both treatments have significant disadvantages. These types of treatment carry the risk of transferring disease from animals and/or humans to the patient; there is also a risk of host local allergic reaction. Bone substitutes are devoid of the above risks and therefore they could be used alternatively to xenografts and allografts. GreenBone is a ceramic resorbable bone scaffold that has very similar structure to bone. It can be produced in large quantities, shaped easily and sterilised without losing its properties. Consequently, it is an ideal substitute that could be used to fill bone defects. This study will assess the safety of using GreenBone treatment of long bone defects up to 6 cm. Moreover it will assess its capacity of promoting new bone formation. The investigators will recruit 25 patients with long bone defect and instead of bovine xenograft we will use the GreenBone implant for the long bone reconstruction. Patients will be followed up for 12 months in total.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female Patients.
2. Patients aged ≥ 18 and ≤ 65 years old.
3. Patients requiring long bone defect reconstructions up to 3 cm, resulting from high-energy traumatic events, or from the treatment of complex bone non-unions in the extremities (arms and legs), or patients undergoing the second stage of the Masquelet technique.
4. Patients understanding the nature of the study and providing their informed consent to participation.
5. Patients willing and able to attend the follow-up visits and procedures foreseen by study protocol.

Please note: after interim analysis review by the DSMB, inclusion criteria n. 3 will be modified as follows (all Investigators will be notified by the Sponsor, and adequate training by Clinical Research Associate-CRA will be conducted):

Change of inclusion criteria n. 3: Patients requiring long bone defect reconstructions longer than 3 cm and up to 6 cm, resulting from high-energy traumatic events, or from the treatment of complex bone non-unions in the extremities (arms and legs), or patients undergoing the second stage of the Masquelet technique.

Exclusion Criteria:

1. Patients with bone infection at the time of enrolment.
2. Patients with bone malignant tumor(s) at the time of enrolment.
3. Patients who have been treated with chemotherapy or radiotherapy within 12 months before the enrolment.
4. Patients with concomitant infectious systemic diseases at the time of enrolment.
5. Patients with known inflammatory systemic diseases at the time of enrolment.
6. Patients with concomitant myeloproliferative disorders at the time of enrolment.
7. Patients currently treated with systemic immunosuppressive agents, excluding steroids.
8. Patients with active autoimmune disease.
9. Patients with a pre-existing calcium metabolism disorder (i.e. hypercalcemia).
10. Known hyperthyroidism or autonomous thyroid adenoma.
11. Patients with coagulopathy or bleeding disorders.
12. Patients who are not allowed to undergo the study procedures involving imaging (X-rays, CT scan) based on Investigator's judgement.
13. Patients with known or suspected allergy or hypersensitivity to the GreenBone Implant components.
14. Patients who are participating or have participated in other clinical studies within the 30 days before the study enrolment.
15. Patients identified by the Investigator to have intra-operative findings that may preclude conduct of study procedure.
16. Patients with occurrence of major intra-operative complications that require resuscitation or deviation from the planned surgical procedure.
17. Women who are pregnant or breast-feeding or who wish to become pregnant during the period of the clinical investigation and for three months later.
18. Female Patients of childbearing age (less than 24 months after the last menstrual cycle) who do not use adequate contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Giannoudis, MD, Principal Investigator — Leeds Teaching Hospital NHS
Locations (8):
- Orthopedic and Traumatology Clinic, University Clinical Center of Republic of Srpska, Banja Luka, Republika Srpska, Bosnia and Herzegovina
- Orthopedic Surgery Section, Division of Surgery,Rambam Health Care Campus, Haifa, Israel
- Italy (3):
  - UOC di Ortopedia e Traumatologia - Ospedali Civili di Brescia, Brescia, Lombardy
  - Unitá Operativa di Traumatologia,Humanitas Research Hospital, Rozzano, Milano
  - U.O.C. Ortopedia e Traumatologia - Osp. Maggiore "C.A. Pizzardi", Bologna
- Orthopedic Surgery Section, Global Care Surgery Hospital, Novi Sad, Serbia
- Clinical Department for Traumatology,University Medical Center of Ljubljana, Ljubljana, Slovenia
- Department of Trauma and Orthopaedic Surgery, Leeds General Infirmary, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment phase started in January 2019
Groups:
- Surgical Repair of Long Bone Defects: The Patients in the study group will be surgically treated and the GreenBone Bone Substitute will be implanted
  surgical repair of long bone defects: Current treatment of bone defects usually implies the use of bone grafts and/or biocompatible materials, to create a scaffold that bridges the defect, favoring the migration of cells from the neighboring tissues to fill the gap. Autograft and Allograft are the treatments most currently used for large bone loss, but both treatments have significant disadvantages. Different types of synthetic materials have been tested for repair of long bone gaps.
  However, at the moment, there is not any bone substitute with the ideal/desirable osteoinductive, osteoconductive and mechanical properties. GreenBone Implant is a synthetic, acellular, reabsorbable, new generation bone graft, being suitable for surgical reconstruction of bone defects.
Period: Overall Study
Arm/Group | Surgical Repair of Long Bone Defects
Started | 16
Completed | 11
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: Only patients treated for bone defect repair were included in the analysis population (16 participants).
Arm/Group | Surgical Repair of Long Bone Defects
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants] — Population: Only patients treated for bone defect repair were included in the analysis population (16 participants)
  Participants
    <=18 years | 0
    Between 18 and 65 years | 15
    >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only patients treated for bone defect repair were included in the analysis population (16 participants)
  Participants
    Female | 4
    Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only patients treated for bone defect repair were included in the analysis population (16 participants)
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 1
    White | 15
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Population: Only patients treated for bone defect repair were included in the analysis population (16 participants)
  participants
    Italy | 9
    United Kingdom | 1
    Israel | 1
    Serbia | 4
    Bosnia and Herzegovina | 1
Bone defect dimension [Mean (Standard Deviation); unit: cm] — Treatment of bone defects up to 3 cm
  cm | 2.3 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Evaluation of adverse events rate during the study period.
Time Frame: Overall study period up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Repair of Long Bone Defects
Number analyzed (Participants) | 16
Participants | 16
Statistical Analysis 1: Comparison: Surgical Repair of Long Bone Defects; Test type: Other — Descriptive statistical analysis; Descriptive statistical analysis

2. Secondary Outcome: Bone Union (Bone Healing) Evaluation Through Modified Lane and Sandhu Radiological Scoring System
Description: Evaluation of the bone regeneration in the area of intervention in comparison to baseline (V1), by means of X-ray and/or CT scan examination, on visits V3, V4, V5, V6, V7 and V8. X-ray scoring systems have been implemented according to the criteria proposed by modified Lane and Sandhu Radiological Scoring System (Lane 1987). This scoring system evaluates bone formation and union. To evaluate the bone formation, there is a scale with 5 points, from 0 to 4 (0=No evidence of bone formation-4=Bone formation occupying 100% of defect). To evaluate bone union, there is a scale with 3 points, from 0 to 2 (0=Non-union-2=Radiographic union).
Time Frame: At the end of visits 1,3,4,5,6,7,8 (respectively performed at screening and 1,2,3,6,9,12 months after the surgery, each visit is 1 day)
Population: Patients that achieved the complete follow-up up to 12 months (11 out of the 16 patients)
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Repair of Long Bone Defects
Number analyzed (Participants) | 11
Participants
  Bone union (Bone healing) | 7
  Possible bone union (Possible healing) | 3
  Not union (not healing) | 1

3. Secondary Outcome: Bone Regeneration Evaluation Through Modified Lane and Sandhu Radiological Scoring System
Description: as for outcome 2
Time Frame: as for outcome 2
Population: Patients that achieved the complete follow-up up to 12 months (11 out of the 16 patients)
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Repair of Long Bone Defects
Number analyzed (Participants) | 11
Participants
  Bone formation occupying 100% of defect | 4
  Bone formation occupying 75% of defect | 3
  Bone formation occupying 50% of defect | 4

4. Secondary Outcome: Evaluation of Pain
Description: Evaluation of degree of pain perceived by the Patient, by means of a Visual Analogue Score (VAS/0-10 point scale), on visits V1, V3, V4, V5, V6, V7 and V8. The Visual Analogue Score (VAS) that a scale with 10 points, from 0 to 10, 0 indicates "no pain at all" and 10 the "worst pain ever".
Time Frame: as for outcome 2
Population: Patients surgically treated with GreenBone Bone Substitute and that completed all follow-up visits
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Surgical Repair of Long Bone Defects
Number analyzed (Participants) | 16
score on a scale
  VAS score - visit 1 | 5.38 (2.25)
  VAS score - visit 3: number analyzed (Participants) | 15
  VAS score - visit 3 | 3.47 (1.85)
  VAS score - visit 4: number analyzed (Participants) | 13
  VAS score - visit 4 | 2.92 (1.61)
  VAS score - visit 5: number analyzed (Participants) | 14
  VAS score - visit 5 | 3.29 (1.33)
  VAS score - visit 6: number analyzed (Participants) | 13
  VAS score - visit 6 | 2.46 (1.71)
  VAS score - visit 7: number analyzed (Participants) | 10
  VAS score - visit 7 | 2.8 (2.15)
  VAS score - visit 8: number analyzed (Participants) | 11
  VAS score - visit 8 | 2.27 (2.28)

5. Secondary Outcome: Evaluation of Quality-of-Life
Description: Evaluation of Quality-of-Life by means of EuroQoL EQ-5D-5L Validated Questionnaire, on visits V1, V3, V4, V5, V6, V7 and V8. The EQ-5D-5L is a descriptive system. This system comprises the same 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems.
Time Frame: as for outcome 2
Reporting Status: Not Posted

6. Secondary Outcome: Global Tolerability of Patient to Treatment
Description: Evaluation of global tolerability to treatment of Patient (by the Investigator), through a standardized questionnaire, on visits V3, V4, V5, V6, V7 and V8. Global Tolerability Questionnaire is a questionnaire with 6 questions that are completed by the investigator in order to evaluate the operated site.
Time Frame: At the end of visits 3,4,5,6,7,8 (respectively performed 1,2,3,6,9,12 months after the surgery, each visit is 1 day)
Reporting Status: Not Posted

7. Secondary Outcome: Reinterventions Number
Description: Evaluation of the number of re-interventions occurring for the Patient throughout the 12-month observation period.
Time Frame: between 1 and 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Description: An adverse event (AE) is defined as any untoward medical occurrence, unintended disease or injury or any untoward clinical signs (including an abnormal laboratory finding) in subjects, users or other persons whether or not related to the investigational medical device.
Arm/Group | Surgical Repair of Long Bone Defects
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 8/16
Other Adverse Events (participants affected / at risk) | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgical Repair of Long Bone Defects (N=16)
Fixation system breakage (Surgical and medical procedures) | 5 (5) — SAE not related to GreenBone implant.
Fracture non-union (Surgical and medical procedures) | 1 (1) — SAE not related to GreenBone implant.
Open reduction with external fixation (Surgical and medical procedures) | 1 (1) — SAE not related to GreenBone implant.
Pseudarthrosis (Surgical and medical procedures) | 1 (1) — SAE not related to GreenBone implant.
Muscle abscess (Skin and subcutaneous tissue disorders) | 1 (1) — SAE not related to GreenBone implant.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgical Repair of Long Bone Defects (N=16)
Allergic Reaction (Musculoskeletal and connective tissue disorders) | 1 (1)
External fixator loosening (Surgical and medical procedures) | 1 (1)
Wound dehiscence (Musculoskeletal and connective tissue disorders) | 1 (1)
Itching (Musculoskeletal and connective tissue disorders) | 1 (1)
Occasional serous drainage (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in leg or arm (Musculoskeletal and connective tissue disorders) | 3 (7)
Joint instability (Musculoskeletal and connective tissue disorders) | 1 (1)
Artery rupture (Injury, poisoning and procedural complications) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2)
Presbyopia (Eye disorders) | 1 (1)
Rectal pain (Eye disorders) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/90/NCT03884790/Prot_SAP_000.pdf